CLINICAL TRIAL: NCT05351606
Title: Integrating Tobacco Use Cessation Into HIV Care and Treatment in Ministry of Health Facilities in Kisumu County, Kenya
Brief Title: Integrating Tobacco Use Cessation Into HIV Care and Treatment in Kisumu County, Kenya
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kenya Medical Research Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22639; 1U01CA261620-01 (NIH)
Record Dates: First submitted 2022-02-16; First posted 2022-04-28 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Tobacco Use Cessation; Tobacco Use
Keywords: Integrated Education; Behavioral Counselling; Nicotine Replacement therapy
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use | interventions — Bupropion; Tobacco Use Cessation Devices; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Brief Intervention (Experimental): Participants will receive one time tobacco use cessation counseling and quitline number.
  Interventions: Behavioral: Tobacco Use Cessation Counselling Sessions
- Intensive Intervention (Experimental): Participants will receive intensive behavioral counseling spread over 12 sessions, Nicotine Replacement Therapy and Bupropion, and the quitline number.
  Interventions: Behavioral: Tobacco Use Cessation Counselling Sessions; Drug: Bupropion; Drug: Nicotine patch; Drug: Nicotine lozenge
- Cross-over Intervention (Experimental): Participants in the brief arm who are still using tobacco at the end of twelve months were invited to participate in a cross-over study whereby they would, if eligible, would receive the intensive intervention.
  Interventions: Behavioral: Tobacco Use Cessation Counselling Sessions; Drug: Bupropion; Drug: Nicotine patch; Drug: Nicotine lozenge

INTERVENTIONS:
Behavioral: Tobacco Use Cessation Counselling Sessions — Counseling sessions will be given in person
Drug: Bupropion — Given orally
  Other Names: Wellbutrin; Zyban
  Arms: Cross-over Intervention; Intensive Intervention
Drug: Nicotine patch — Given transdermally
  Other Names: Nicotine Replacement Therapy (NRT)
  Arms: Cross-over Intervention; Intensive Intervention
Drug: Nicotine lozenge — Given orally
  Other Names: Nicotine lozenge product; NRT
  Arms: Cross-over Intervention; Intensive Intervention

SUMMARY:
People living with HIV (PLHIV) have higher rates of tobacco use than the general population and higher rates of disease and death compared with PLHIV who do not use tobacco. This project will evaluate the impact of integrating an intensive tobacco use cessation intervention compared to a brief intervention within HIV care clinics in Kisumu County, Kenya.

There is evidence that PLHIV in Africa are more likely to use tobacco than the general population. Kenya is an example of a country coping with the dual epidemic of HIV and tobacco, with an estimated 1.5 million PLHIV and 2.5 million tobacco users. HIV remains one of the country's leading causes of morbidity and mortality, with an estimated 46,000 adults acquired HIV and 25,000 persons died of HIV in 2018. Tobacco use among the general population is estimated to be 11.6% (19.1% among men and 4.5% among women). The impact of tobacco use among PLHIV in Kenya has yet to be fully understood. There has been no research or initiatives in Kenya to support PLHIV to quit tobacco use in a primary care setting, a gap that this study seeks to address. In 2017, Kenya's Ministry of Health launched the National Guidelines for Tobacco Dependence Treatment and Cessation. This project will also examine the integration of the Guidelines' interventions into Ministry of Health HIV care clinics in Kisumu County.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the success of the intensive versus a brief smoking cessation intervention after one year.

SECONDARY OBJECTIVES:

I. To examine the success of the intensive versus a brief smoking cessation intervention at 1 month, 3 months and 6 months.

II. To compare the HIV viral load with abstinence rates for each of the interventions.

STUDY OVERVIEW:

The investigator will conduct a cluster randomized controlled trial at 20 Ministry of Health HIV clinics in Kisumu Kenya, recruiting 580 patients who will be randomized to one of 2 conditions to investigate the effectiveness of an intensive versus a brief intervention aimed at smoking cessation.

Participants will be assessed at baseline, one month, three months, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Human immunodeficiency virus (HIV)-seropositive,
* Age >=18 years
* Currently taking or initiating antiretroviral therapy (ART)
* Access to mobile phone for phone or text follow up visit (intensive intervention only)
* Able to read or be read short message service (SMS) messages (intensive intervention only).

Tobacco inclusion criteria:

* Current tobacco users, who have used tobacco in the past 7 days;
* Must have smoked at least 100 cigarettes in lifetime, and at least 5 cigarettes per day biochemically verified by expired Carbon Monoxide (CO) >= 5-6 parts per million (ppm).

Exclusion Criteria:

* Advanced HIV disease, age < 18 years
* Unable to provide verbal informed consent
* Unwilling to be contacted by clinic for follow up

Additional exclusion criteria in the intensive intervention group:

* Myocardial Infarction (MI) in the 2 weeks prior to signing consent
* Pregnant (NRT and Bupropion may be contraindicated).
* Patients for whom Bupropion is contraindicated (e.g. history of seizures, recent use of Monoamine oxidase (MAO) inhibitors, breastfeeding, and whose ART protocol present, as per prescription guidance, contraindications).
* Prior disclosure of HIV status to the phone owner for those who use phones will be required to prevent inadvertent disclosure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who have abstained from tobacco use at 12 months | 12 months
  The point prevalent abstinence rate will be reported as the proportion of participants who have abstained from tobacco use and will be dichotomized as either smoking or abstinent. Abstinence is determined by a self-report of 7-day continuous abstinence verified by a salivary cotinine test.

SECONDARY OUTCOMES:
Proportion of participants who have abstained from tobacco use at 1 month | 1 month
  The point prevalent abstinence rate will be reported as the proportion of participants who have abstained from tobacco use and will be dichotomized as either smoking or abstinent. Abstinence is determined by a self-report of 7-day continuous abstinence verified by a expired carbon monoxide reading of less than 5 parts per million (ppm).
Proportion of participants who have abstained from tobacco use at 3 months | 3 months
  The point prevalent abstinence rate will be reported as the proportion of participants who have abstained from tobacco use and will be dichotomized as either smoking or abstinent. Abstinence is determined by a self-report of 7-day continuous abstinence verified by a expired carbon monoxide reading of less than 5 parts per million (ppm).
Proportion of participants who have abstained from tobacco use at 6 months | 6 months
  The point prevalent abstinence rate will be reported as the proportion of participants who have abstained from tobacco use and will be dichotomized as either smoking or abstinent. Abstinence is determined by a self-report of 7-day continuous abstinence verified by a salivary cotinine test.
Median HIV Viral load by abstinence status | 12 months
  Routine viral load measurement will be taken from the participants at the 12 month visit and the median viral load in copies per ml will be reported along with the interquartile range (IQR) by biochemically verified abstinence status for each group at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Bialous, Dr PH, Principal Investigator — University of California, San Francisco
Locations (1):
- Kenya Medical Research Institute (KEMRI), Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No